CLINICAL TRIAL: NCT01057121
Title: A Phase I/II Study of Lenalidomide in Patients With AIDS-Associated Kaposi's Sarcoma
Brief Title: Lenalidomide in Treating Patients With AIDS-Associated Kaposi's Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02923; NCI-2012-02923 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000664131; AMC-070 (Other: AIDS - Associated Malignancies Clinical Trials Consortium); AMC-070 (Other: CTEP); U01CA121947 (NIH)
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: AIDS-Related Kaposi Sarcoma; Recurrent Kaposi Sarcoma
Keywords: HIV Infections
MeSH Terms: conditions — AIDS-related Kaposi sarcoma; Sarcoma, Kaposi; HIV Infections | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Patients receive lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles. Sequential cohorts were entered at 10 mg/day, 15 mg/day, 20 mg/day and 25 mg/day using a 3+3 design to determine the MTD
  Other Names: Revlimid

SUMMARY:
This phase I/II trial studies the side effects and best dose of lenalidomide and to see how well it works in treating patients with acquired immunodeficiency syndrome (AIDS)-related Kaposi sarcoma (KS). Lenalidomide may stop the growth of tumor cells by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of single agent lenalidomide in subjects with AIDS-related KS. (Phase I) II. Evaluate the overall clinical response of KS tumors to lenalidomide with subset assessments of partial response (PR) and complete response (CR). (Phase II)

SECONDARY OBJECTIVES:

I. Evaluate the effect of lenalidomide on human immunodeficiency virus (HIV) plasma viral loads.

II. Determine the effects of lenalidomide on T-lymphocyte subsets, including natural killer (NK) cells.

III. Evaluation of time to response, time to relapse, and time to death amongst subjects receiving lenalidomide.

IV. Determine the effect of lenalidomide on human herpesvirus (HHV)-8. V. Assess lenalidomide effects on HHV-8 copy number in peripheral blood mononuclear cell (PBMC), and plasma and whether changes in viral copy number measured in PBMC or plasma are associated with clinical response of KS tumors.

VI. Monitor HHV-8 gene expression in KS biopsy specimens and PBMC pre- and post-lenalidomide and assess whether changes in viral gene expression in tumor biopsy are associated with clinical response.

VII. Assess whether changes in viral copy number in the compartments assayed occur in concert or independently with changes in viral antigen expression in biopsy specimens.

VIII. Assess effects of lenalidomide on growth factors relevant to tumor proliferation (i.e., interleukin [IL]-1beta, IL-2, IL-4, IL-5, IL-6, IL-10, IL-15, IL-12p70, tumour necrosis factor [TNF]alpha, and interferon gamma [IFN]gamma).

IX. Characterize the effects of lenalidomide on viral and cellular gene in KS tumor biopsies.

X. Assess changes in NK cell number (PBMC and tumor) and function pre- and post-lenalidomide.

XI. Assess the sensitivity and specificity of dermal adhesive strip samples to detect KS and the effects of lenalidomide on the lesions.

OUTLINE: This is a multicenter study. This is a phase I, dose-escalation study of lenalidomide followed by a phase II study.

Patients receive lenalidomide orally (PO) once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven KS involving skin with or without visceral involvement either newly diagnosed or refractory to or intolerant of one or more prior therapies
* Patients must have cutaneous lesion(s) amenable to four 3 mm tumor biopsies during the study (either 4 separate lesions measuring > 4 mm each OR 2 separate lesions measuring > 8 mm each) and at least five additional lesions measurable for assessment with no improvement over the past month
* Serologic documentation of HIV infection by any of the Food and Drug Administration (FDA)-approved tests
* Karnofsky performance status >= 60%
* Hemoglobin >= 8 g/dL
* Absolute neutrophil count (ANC) >= 1,000 cells/mm^3
* Platelet count >= 100,000/mm^3
* Calculated (method of Cockcroft-Gault) creatinine clearance (CrCl) >= 60 mL/min in the Phase I and CrCl >= 30 mL/min in the Phase II (creatinine clearance may also be obtained by the 24-hour collection method at the investigator's discretion)
* Total bilirubin should be =< 1.5x upper limit of normal (ULN); if, however, the elevated bilirubin is felt to be secondary to Atazanavir therapy, patients will be allowed to enroll on protocol if the total bilirubin is =< 3.5 mg/dL provided that the direct bilirubin is normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3x ULN
* Life expectancy >= 3 months
* Ability and willingness to give informed consent
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours prior to starting Cycle 1 of lenalidomide; further, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide, during receipt of lenalidomide, and 28 days after discontinuation of lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure
* Patients must, in the opinion of the investigator, be capable of complying with the protocol
* All patients must be on antiretroviral therapy for HIV infection with CD4 count > 50/mm^3 and viral load < 2,000 copies/mL; patients must be on a stable regimen for at least 12 weeks prior to study entry; patients may receive any FDA approved antiretroviral therapy except for zidovudine

  * There should be no evidence for improvement in KS in the 3 months prior to study entry, unless there is evidence for progression of KS in the 4 weeks immediately prior to study entry
  * If antiretroviral regimen contains zidovudine and viral load is suppressed (as measured by HIV viral load =< 200/mL), then antiretroviral therapy must be adjusted to a less toxic therapy not containing zidovudine and enrollment may proceed without waiting 12 weeks; if on zidovudine-containing therapy and viral load is not suppressed (as measured by HIV viral load >= 200/mL), then antiretroviral therapy must be adjusted to a less toxic regimen allowing for optimal viral suppression and must demonstrate stability for at least 12 weeks prior to study entry
* Patients with any history of pulmonary embolism (PE) or deep venous thrombosis (DVT) or predisposing clotting risk factors must be on anticoagulation at therapeutic dosing

Exclusion Criteria:

* Concurrent, acute, active opportunistic infection other than oral thrush or genital herpes within 14 days of enrollment
* Patients for whom front-line cytotoxic therapy is indicated (i.e. symptomatic visceral or pulmonary KS or symptomatic KS impairing functional status)
* Concurrent neoplasia requiring cytotoxic therapy
* Acute treatment for an infection (other than oral thrush or genital herpes) or other serious medical illness within 14 days of study entry
* Anti-neoplastic treatment for KS (including chemotherapy, radiation therapy, local therapy including topical 5-FU, biological therapy, or investigational therapy) within four weeks of study entry
* Any steroid treatment except for that required for replacement therapy in adrenal insufficiency or inhaled steroids for the treatment of asthma
* Patient is =< 2 years free of another primary malignancy; exceptions include the following:

  * Basal cell skin cancer
  * Cervical carcinoma in situ
  * Anal carcinoma in situ
* Previous local therapy of any KS-indicator lesion unless the lesion has clearly progressed since treatment; any prior local treatment to indicator lesions regardless of the elapsed time should not be allowed unless there is evidence of clear-cut progression of said lesion
* Use of any investigational drug or treatment within 4 weeks prior to enrollment
* Physical or psychiatric conditions that in the estimation of the investigator place the patient at high risk of toxicity or non-compliance
* Female patients who are pregnant or breast-feeding
* Patients with a history of DVT or PE within 1 year
* Patients requiring blood transfusions to maintain Hgb eligibility
* Patients on erythropoietin-stimulating agents (ESA) unless also on therapeutic anticoagulation
* Patients with CD4 < 50 mm^3 and/or viral load > 2,000 copies/mL
* Patients on estrogen therapy unless also on therapeutic anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-08-27 (Actual); Primary Completion 2014-08-04 (Actual); Study Completion 2014-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Shimabukuro, Principal Investigator — AIDS Associated Malignancies Clinical Trials Consortium
Locations (13):
- United States (13):
  - UCLA Center for Clinical AIDS Research and Education, Los Angeles, California
  - University of California San Diego, San Diego, California
  - San Francisco General Hospital, San Francisco, California
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Cancer Center of Hawaii-Hawaii AIDS Clinical Research Program, Honolulu, Hawaii
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Thomas Street Clinic, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Reid EG, Shimabukuro K, Moore P, Ambinder RF, Bui JD, Han S, Martinez-Maza O, Dittmer DP, Aboulafia D, Chiao EY, Maurer T, Baiocchi R, Mitsuyasu R, Wachsman W; AIDS Malignancy Consortium (AMC). AMC-070: Lenalidomide Is Safe and Effective in HIV-Associated Kaposi Sarcoma. Clin Cancer Res. 2022 Jun 13;28(12):2646-2656. doi: 10.1158/1078-0432.CCR-21-0645. PMID 35247913

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Treatment (Lenalidomide) , 10 mg/Day: Patients receive 10 mg lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
- Phase I: Treatment (Lenalidomide), 15 mg/Day: Patients receive 15 mg lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
- Phase I, Treatment Ienalidomide), 20 mg/Day: Patients receive 20 mg lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
- Phase I: Treatment (Lenalidomide), 25 mg/Day; Phase II: Treatment (Lenalidomide), 25 mg/Day: Patients receive 25 mg lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Period: Phase I: 10 mg/Day Lenalidomide
Arm/Group | Phase I: Treatment (Lenalidomide) , 10 mg/Day | Phase I: Treatment (Lenalidomide), 15 mg/Day | Phase I, Treatment Ienalidomide), 20 mg/Day | Phase I: Treatment (Lenalidomide), 25 mg/Day | Phase II: Treatment (Lenalidomide), 25 mg/Day
Started | 3 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Phase I: 15 mg/Day Lenolidomide
Arm/Group | Phase I: Treatment (Lenalidomide) , 10 mg/Day | Phase I: Treatment (Lenalidomide), 15 mg/Day | Phase I, Treatment Ienalidomide), 20 mg/Day | Phase I: Treatment (Lenalidomide), 25 mg/Day | Phase II: Treatment (Lenalidomide), 25 mg/Day
Started | 0 | 3 | 0 | 0 | 0
Completed | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Phase I: 20 mg/Day Lenalidomide
Arm/Group | Phase I: Treatment (Lenalidomide) , 10 mg/Day | Phase I: Treatment (Lenalidomide), 15 mg/Day | Phase I, Treatment Ienalidomide), 20 mg/Day | Phase I: Treatment (Lenalidomide), 25 mg/Day | Phase II: Treatment (Lenalidomide), 25 mg/Day
Started | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Phase I: 25 mg/Day Lenalidomide
Arm/Group | Phase I: Treatment (Lenalidomide) , 10 mg/Day | Phase I: Treatment (Lenalidomide), 15 mg/Day | Phase I, Treatment Ienalidomide), 20 mg/Day | Phase I: Treatment (Lenalidomide), 25 mg/Day | Phase II: Treatment (Lenalidomide), 25 mg/Day
Started | 0 | 0 | 0 | 6 | 0
Completed | 0 | 0 | 0 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Phase II: 25 mg/Day Lenalidomide
Arm/Group | Phase I: Treatment (Lenalidomide) , 10 mg/Day | Phase I: Treatment (Lenalidomide), 15 mg/Day | Phase I, Treatment Ienalidomide), 20 mg/Day | Phase I: Treatment (Lenalidomide), 25 mg/Day | Phase II: Treatment (Lenalidomide), 25 mg/Day
Started | 0 | 0 | 0 | 0 | 23
Completed | 0 | 0 | 0 | 0 | 23
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I - Treatment (Lenalidomide); Phase II - Treatment (Lenalidomide): Patients receive lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
- Total: Total of all reporting groups
Arm/Group | Phase I - Treatment (Lenalidomide) | Phase II - Treatment (Lenalidomide) | Total
Number analyzed (Participants) | 15 | 23 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (11.8) | 46.9 (8.2) | 47.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 23 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 11 | 18 | 29
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 1 | 5 | 6
  White | 12 | 14 | 26
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 23 | 38

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Lenalidomide Defined as the Dose Level at Which 0/6 or 1/6 Subjects Experience Dose Limiting Toxicity (DLT) With the Next Higher Dose Having at Least 2/3 or 2/6 Subjects Encountering DLT (Phase I)
Description: Maximum tolerated dose (MTD) of lenalidomide defined as the dose level at which 0/6 or 1/6 subjects experience dose limiting toxicity (DLT) with the next higher dose having at least 2/3 or 2/6 subjects encountering DLT (Phase I). Toxicities will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. Using a 3+3 design, the MTD is defined as the level at which 0/6 or 1/6 patients experiences at dose-limiting toxicity in the first cycle.
Time Frame: 28 days
Population: Only patients in the phase I portion of the study were evaluated for this outcome measure.
Measure: Number; unit: mg per day of lenalidomide
Groups:
- Phase I - Treatment (Lenalidomide): Phase I: Patients receive lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles This arm includes patients treated at the 10 mg/day dose (N=3), 15 mg/day dose (N=3), 20 mg/day dose (N=3) and 25 mg/day dose (N=6)
Arm/Group | Phase I - Treatment (Lenalidomide)
Number analyzed (Participants) | 15
mg per day of lenalidomide | 25

2. Primary Outcome: Tumor Response Rate
Description: Percentage of patients who achieve a partial or complete response Complete response was defined as the absence of any detectable residual disease, including tumor-associated edema, that persisted for at least 4 weeks.
  Partial response was defined as no new lesions (skin or oral), or new visceral sites of involvement (or the appearance or worsening of tumor-associated edema or effusions), and a 50% or greater decrease in the number of all previously existing lesions that lasted for at least 4 weeks, or complete flattening of at least 50% of all previously raised lesions, or a 50% or greater decrease in the sum of the products of the largest perpendicular diameters of the marker lesions.
Time Frame: Up to 30 days after completion of study treatment
Population: Patients who were evaluable for response. To be evaluable for response, the patient had to complete at least one cycle of treatment.
Measure: Number (95% Confidence Interval); unit: percent of participants who responded
Groups:
- Phase I - 10 mg/Day (Lenalidomide): Patients received 10 mg/day lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
- Phase I - 15 mg/Day (Lenalidomide): Patients received 15 mg/day lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
- Phase I: 20 mg/Day Lenalidomide: Patients received 20 mg/day lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
- Phase I: 25 mg/Day Lenalidomide; Phase II: 25 mg/Day Lenalidomide: Patients received 25 mg/day lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
Arm/Group | Phase I - 10 mg/Day (Lenalidomide) | Phase I - 15 mg/Day (Lenalidomide) | Phase I: 20 mg/Day Lenalidomide | Phase I: 25 mg/Day Lenalidomide | Phase II: 25 mg/Day Lenalidomide
Number analyzed (Participants) | 3 | 3 | 2 | 5 | 19
percent of participants who responded | 0 [0 to 0] | 0 [0 to 0] | 50 [1 to 99] | 80 [28 to 99] | 53 [30 to 75]

3. Secondary Outcome: Time to Death
Description: Percentage of patients who died
Time Frame: Up to 30 days after completion of study treatment
Population: Study participants who died on study.
Measure: Number; unit: percentage of participants who died
Groups:
- Phase I - 10 mg/Day Lenalidomide: Patients received 10 mg/day lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
- Phase I - 15 mg/Day Lenalidomide: Patients received lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
Arm/Group | Phase I - 10 mg/Day Lenalidomide | Phase I - 15 mg/Day Lenalidomide | Phase I: 20 mg/Day Lenalidomide | Phase I: 25 mg/Day Lenalidomide | Phase II: 25 mg/Day Lenalidomide
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 23
percentage of participants who died | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Time to Relapse
Description: Percentage of participants who relapsed
Time Frame: Up to 30 days after completion of study treatment
Population: Patients who relapsed
Groups:
- Phase I - 10 mg/Day Treatment (Lenalidomide): Patients receive 10 mg/day of lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
- Phase I - 15 mg/Dah Treatment (Lenalidomide): Patients receive 15 mg/day lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
- Phase I - 20 mg/Day Treatment (Lenalidomide): Patients receive 20 mg/day lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
- Phase I: Treatment (Lenalidomide), 25 mg/Day; Phase II: 25 m/Day Treatment (Lenalidomide): Patients receive 25 mg/day lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
Arm/Group | Phase I - 10 mg/Day Treatment (Lenalidomide) | Phase I - 15 mg/Dah Treatment (Lenalidomide) | Phase I - 20 mg/Day Treatment (Lenalidomide) | Phase I: Treatment (Lenalidomide), 25 mg/Day | Phase II: 25 m/Day Treatment (Lenalidomide)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Time to Response
Description: time from enrollment to first response (complete or partial) as defined below: Complete response is defined as the absence of any detectable residual disease, including tumor-associated edema, persisting for at least 4 weeks.
  Partial response is defined as no new lesions (skin or oral), or new visceral sites of involvement (or the appearance or worsening of tumor-associated edema or effusions), and a 50% or greater decrease in the number of all previously existing lesions lasting for at least 4 weeks, or complete flattening of at least 50% of all previously raised lesions, or a 50% or greater decrease in the sum of the products of the largest perpendicular diameters of the marker lesions.
Time Frame: Up to 30 days after completion of study treatment
Population: Participants who had a complete or partial responses
Measure: Median (Full Range); unit: weeks
Groups:
- Phase I - 10 mg/Day Treatment (Lenalidomide): Patients receive 10 mg/day lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
- Phase I: 20 mg/Day Treatment (Lenalidomide): Patients receive 20 mg/day lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
- Phase I: 25 mg/Day Treatment (Lenalidomide); Phase II: 25 m/Day Treatment (Lenalidomide): Patients receive 25 mg/day lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
Arm/Group | Phase I - 10 mg/Day Treatment (Lenalidomide) | Phase I - 15 mg/Dah Treatment (Lenalidomide) | Phase I: 20 mg/Day Treatment (Lenalidomide) | Phase I: 25 mg/Day Treatment (Lenalidomide) | Phase II: 25 m/Day Treatment (Lenalidomide)
Number analyzed (Participants) | 0 | 0 | 1 | 4 | 10
weeks |  |  | 8 [8 to 8] | 20.5 [12 to 28] | 13 [4 to 38]

6. Other Pre Specified Outcome: Relationship Between Clinical Response and Quantitative Measures of Kaposi's Sarcoma-associated Herpesvirus (KSHV)/HHV-8 and HIV Viral Load
Description: Spearman rank correlation analysis will be used to evaluate the relationship between the qualification of baseline KSHV/HHV-8, HIV viral load and time to progression, and response duration.
Time Frame: Up to 30 days after completion of study treatment
Population: The KSHV (HHV-8) assays were run, but the results were unreliable.
Arm/Group | Phase I - Treatment (Lenalidomide) | Phase II - Treatment (Lenalidomide)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Phase I: 10 mg/Day Lenalidomide: Patients receive 10 mg lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
- Phase I: 15 mg/Day Lenalidomide: Patients receive 15 mg lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
- Phase I: 20 mg/Day Lenalidomide: Patients receive 20 mg lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
- Phase I and II: 25 mg/Day Lenalidomide: Patients receive 25 mg lenalidomide PO once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Lenalidomide: Lenalidomide is administered daily on days 1-21 of a 28-day cycle. The maximum duration of treatment is 12 28-day cycles
Arm/Group | Phase I: 10 mg/Day Lenalidomide | Phase I: 15 mg/Day Lenalidomide | Phase I: 20 mg/Day Lenalidomide | Phase I and II: 25 mg/Day Lenalidomide
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 6/29
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: 10 mg/Day Lenalidomide (N=3) | Phase I: 15 mg/Day Lenalidomide (N=3) | Phase I: 20 mg/Day Lenalidomide (N=3) | Phase I and II: 25 mg/Day Lenalidomide (N=29)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 0 | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: 10 mg/Day Lenalidomide (N=3) | Phase I: 15 mg/Day Lenalidomide (N=3) | Phase I: 20 mg/Day Lenalidomide (N=3) | Phase I and II: 25 mg/Day Lenalidomide (N=29)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 | 2 | 7
Blood and Lymphatic disorders, other (Blood and lymphatic system disorders) | 0 (0) | 0 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 (0) | 1 | 0 | 6
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 | 1 | 13
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 | 0 | 2
Gastroesophageal reflux (Gastrointestinal disorders) | 0 (0) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 6
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 | 0 | 4
Edema - limbs (General disorders) | 1 (1) | 0 | 0 | 3
Fatigue (General disorders) | 2 (2) | 0 | 2 | 16
Fever (General disorders) | 0 (0) | 0 | 0 | 4
Pain (General disorders) | 1 (1) | 0 | 0 | 4
Allergic reaction (Immune system disorders) | 1 (1) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 (0) | 0 | 0 | 2
Skin infection (Infections and infestations) | 1 (2) | 0 | 0 | 4
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 | 0 | 4
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 | 0 | 4
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 | 0 | 4
Lymphocyte count decreased (Investigations) | 0 (0) | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 0 (0) | 1 | 2 | 12
Platelet count decreased (Investigations) | 1 (1) | 1 | 0 | 5
Weight loss (Investigations) | 0 (0) | 0 | 1 | 1
White blood cell decreased (Investigations) | 0 (0) | 0 | 1 | 6
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 | 0 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 | 0 | 3
Metaolism and nutrition disorders, other (Metabolism and nutrition disorders) | 2 (2) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 1 | 2
Dizziness (Nervous system disorders) | 0 (0) | 0 | 0 | 4
Headache (Nervous system disorders) | 1 (1) | 0 | 0 | 8
Nervous system disorder, other (Nervous system disorders) | 0 (0) | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 | 0 | 1
Anxiety (Nervous system disorders) | 1 (1) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 (0) | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 0 (0) | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 | 0 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 | 0 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 | 1 | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 | 2 | 10
Skin and subcutaneous tissue disorders, other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 6
Lymphedema (Vascular disorders) | 0 (0) | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 1 (2) | 0 | 0 | 0
Creatinine Increased (Investigations) | 1 (1) | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Investigations, other (Investigations) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less